CLINICAL TRIAL: NCT02188446
Title: Randomised Controlled Multicenter Study.Effect of an Intensive Smoking- and/or Alcohol Cessation Intervention Placed Shortly Before and 5 Weeks After Bladder Cancer Surgery on Postoperative Complications
Brief Title: Intensive Smoking and Alcohol Cessation Intervention in Bladder Cancer Surgery Patients
Acronym: STOP-OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Frederiksberg University Hospital (Other); Aalborg University Hospital (Other); Copenhagen University Hospital at Herlev (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Susanne Vahr lauridsen, MEd, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: F-22841-01
Record Dates: First submitted 2014-05-28; First posted 2014-07-11 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Bladder Cancer; Smoking; Alcohol Consumption
Keywords: Radical cystectomy; Bladder cancer; Smoking cessation; Alcohol cessation; Postoperative complications
MeSH Terms: conditions — Urinary Bladder Neoplasms; Smoking; Alcohol Drinking; Smoking Cessation; Postoperative Complications | interventions — Smoking Devices; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking and alcohol cessation education (Experimental)
  Interventions: Behavioral: Educational programme for smoking and alcohol cessation
- Standard treatment (No Intervention): Standard treatment is information about benefits of stopping drinking and smoking before surgery and if wanted, advice about who to contact to get support.

INTERVENTIONS:
Behavioral: Educational programme for smoking and alcohol cessation — 5 meetings within 6 weeks containing education and pharmacologic support
  Other Names: GSP
  Arms: Smoking and alcohol cessation education

SUMMARY:
Radical cystectomy provides the best cancer-specific survival for muscle-invasive urothelial cancer. However the postoperative morbidity remains at 11-68 %. Smoking and alcohol consumption above two drinks per day is associated with an increased risk of postoperative morbidity. Six-eight weeks of smoking and alcohol abstinence prior to elective surgery is recommended to reduce this risk, but for cancer patients the preoperative period is often very short. This randomised clinical trial (STOP-OP) will reach a conclusion on the effect of a new Gold Standard Programme for both smoking and alcohol cessation Intervention using the Gold Standard Programme (GSP) on the frequency and severity of postoperative complications after bladder cancer surgery.

DETAILED DESCRIPTION:
The study is a multicentre randomised clinical trial involving 110 patients with a risky alcohol intake (exceeding 21 alcohol units (252 g ethanol) per week or/ and daily smoking scheduled for bladder cancer surgery. Patients will be randomised to the 6-weeks GSP or treatment as usual (control). The GSP combines patient education and pharmacologic strategies. The GSP includes benzodiazepine therapy for withdrawal symptoms, controlled disulfiram therapy, and Nicotine replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years scheduled for cystectomy due to bladder cancer
* Daily smoker or/and intake of

  ->21 units (252 g) of alcohol pr week
* Informed consent

Exclusion Criteria:

* Cancelled operation
* Hypersensitivity to benzodiazepines, disulfiram or Nicotine replacement
* Pregnant or breastfeeding women
* Mentally incompetent patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative complications | Up to 6 weeks
  Both number of patients with postoperative complications and number of postoperative complications according to the Clavien Dindo classification will be measured

SECONDARY OUTCOMES:
Postoperative complications | up to 90 days
Smoking and alcohol cessation up to 12 months postoperatively Smoking and alcohol cessation | Up to 12 months postoperatively
Length of stay | From day of surgery to day of discharge
Time to return to work or habitual level of activity | Up to 12 months
Mortality | Up to 12 months postoperatively
Quality of life ( EORTC QLQ BLM 30 and EQ5D) | Up to 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Tønnesen, Professor, Study Chair — WHO-CC, Clinical Health Promotion Centre, Bispebjerg/Frederiksberg University Hospital, DK 2000 Frederiksberg, Denmark
Locations (1):
- Department of Urology, University Hospital of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Merzaai B, Tonnesen H, Rasmussen M, Lauridsen SV. Perioperative Alcohol and Smoking Cessation Intervention: Impact on Other Lifestyles. Semin Oncol Nurs. 2021 Feb;37(1):151116. doi: 10.1016/j.soncn.2020.151116. Epub 2021 Jan 6. PMID 33422365
- [Derived] Lauridsen SV, Thomsen T, Thind P, Tonnesen H. STOP smoking and alcohol drinking before OPeration for bladder cancer (the STOP-OP study), perioperative smoking and alcohol cessation intervention in relation to radical cystectomy: study protocol for a randomised controlled trial. Trials. 2017 Jul 17;18(1):329. doi: 10.1186/s13063-017-2065-6. PMID 28716147
- See also: DaBlaCa study number 6 — http://ducg.dk/dablaca-blaerecancer/forskningsprojekter/